CLINICAL TRIAL: NCT05523037
Title: Comparison of the Effect of Remimazolam With Sevoflurane on Postanesthetic Shivering in Patients Undergoing Laparoscopic Gynecologic Surgery Under General Anesthesia-prospective Observational Study.
Brief Title: Comparison of the Effect of Remimazolam With Sevoflurane on Postanesthetic Shivering
Status: Completed | Type: Observational
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Other Study IDs: WonkwangUH10
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia; Hypothermia
Keywords: shivering; general anesthesia; laparoscopic surgery
MeSH Terms: conditions — Hypothermia | interventions — Sevoflurane; remimazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: Anesthesia induction was achieved by continuous infusion of 6 mg/kg/h of remimazolam, and the maintenance of anesthesia was maintained at a BIS between 40 and 60.
  For the maintenance of anesthesia, the end-tidal concentration of 1 minimum alveolar concentration (MAC) sevoflurane was administered
  Interventions: Drug: Sevoflurane
- Group R: Anesthesia induction was achieved by continuous infusion of 6 mg/kg/h of remimazolam, and the maintenance of anesthesia was maintained at a BIS between 40 and 60.
  For the maintenance of anesthesia, 1-2 mg/kg/h of remimazolam was continuously infused.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Sevoflurane — For the maintenance of anesthesia, the end-tidal concentration of 1 minimum alveolar concentration (MAC) sevoflurane and the concentration was adjusted by 1% stepwise titration
  Groups: Group S
Drug: Remimazolam — For the maintenance of anesthesia, 1-2 mg.kg-1.h-1 of remimazolam was continuously infused.
  Other Names: Byfavo®
  Groups: Group R

SUMMARY:
The incidence of postanesthetic shivering (PAS) after general anesthesia is affected by the anesthesia maintenance agents. This study compared the effect of remimazolam with sevoflurane on PAS in patients with laparoscopic gynecologic surgery under general anesthesia.

DETAILED DESCRIPTION:
Inadvertent perioperative hypothermia and postanesthetic shivering (PAS) are common after anesthesia regardless of anesthesia methods. The incidence of perioperative hypothermia and PAS after general anesthesia has been reported to be 37.5 to 77.2% and 20 to 70%, respectively. Shivering begins when vasoconstriction, a major mechanism to prevent body heat loss, is insufficient. PAS is one of the most common discomforts in the recovery room after general anesthesia. Therefore, PAS is common in hypothermic patients.

Volatile or intravenous anesthetics impair the autonomic thermoregulatory vasoconstriction which usually preserves core body temperature. However, benzodiazepines, such as midazolam, do not significantly impair thermoregulation control, even when used in combination with common opioid doses. Remimazolam, a novel benzodiazepine, has been reported for the thermoregulatory vasoconstriction threshold and onset time of vasoconstriction in terms of core body temperature in patients undergoing robotic-assisted and laparoscopic radical prostatectomy. It decreased the vasoconstriction threshold less than propofol, one of the intravenous anesthetics, and the onset of vasoconstriction was faster than propofol.

Investigators hypothesized that remimazolam reduced the incidence of hypothermia compared to sevoflurane, one of the volatile anesthetics, and eventually lowered the frequency of PAS. Therefore, this study compared the effect of remimazolam with sevoflurane on PAS in patients with laparoscopic gynecologic surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 19 and 65 y, with ASA physical status classes I or II

Exclusion Criteria:

* Patients with history such as thyroid disease, cardiopulmonary disease, blood coagulation disorder, liver dysfunction, cranial nerve disease, alcohol or drug abuse, a known allergy to the study drug, and those who had core body temperature > 38°C or < 36.5°C, BMI > 30 kg.m-2 or febrile illness were excluded. Patients who underwent surgery for less than 60 min, and those who did not consent to this study

Ages: 19 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: patients aged between 19 and 65 y, with ASA physical status classes I or II, who undergoing laparoscopic gynecologic surgery
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
The incidence of postanesthetic shivering (PAS) | during staying in recovery room
  In the recovery room, an attending anesthesiologist observed shivering. The severity of PAS was assessed with a bedside shivering assessment scale, which rated shivering as None (Grade 0): no shivering noted on palpation of the masseter, neck, or chest wall, Mild (Grade 1): shivering localized to the neck and/or thorax only, Moderate (Grade 2): shivering involved gross movement of the upper extremities (in addition to neck and thorax) and Severe (Grade 3): shivering involved gross movements of the trunk and upper and lower extremities

SECONDARY OUTCOMES:
The severity of PAS | during staying in recovery room
  The severity of PAS was assessed with bedside shivering assessment scale, which rate shivering as None (Grade 0): no shivering noted on palpation of the masseter, neck, or chest wall, Mild (Grade 1): shivering localized to the neck and/or thorax only, Moderate (Grade 2): shivering involved gross movement of the upper extremities (in addition to neck and thorax) and Severe (Grade 3): shivering involved gross movements of the trunk and upper and lower extremities
Mean arterial pressure (MAP) | during general anesthesia
  MAP was checked at pre-induction, and after induction, every 10 minutes until the end of surgery.
Heart rate (HR) | during general anesthesia
  HR was checked at pre-induction, and after induction, every 10 minutes until the end of surgery.
Core body temperature | during general anesthesia
  The patient's core body temperature was measured using an infrared tympanic thermometer and the highest temperature among the three measurements was measured before induction of anesthesia and in recovery room. After anesthesia induction, a nasopharyngeal temperature probe was inserted through the nostril to a depth of 9.5 to 10 cm at an appropriate location.

CONTACTS AND LOCATIONS:
Locations (1):
- Wonkwag UH, Iksan, Jeollabukdo, South Korea

IPD SHARING:
Plan to Share IPD: Undecided